CLINICAL TRIAL: NCT06827964
Title: Effects of Nutrition Package (Yingyangbao) Intervention on Children and Adolescents' Health in Myanmar
Brief Title: Practice of Nutrition Package in Myanmar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Ai Zhao, Associate Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THU01-20240170
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Malnutrition in Children
Keywords: Nutrition Package; Malnutrition; Myanmar
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Probiotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Nutrition Package plus Probiotics
  Interventions: Dietary Supplement: Soy-based Nutrition Package; Dietary Supplement: Probiotics
- Group 2 (Experimental): Nutrition package alone
  Interventions: Dietary Supplement: Soy-based Nutrition Package
- Group 3 (No Intervention): Blank control

INTERVENTIONS:
Dietary Supplement: Soy-based Nutrition Package — Dry, vacuum-sealed sachets containing yellow powder, odorless, to be consumed with warm water. Each 12g sachet provides: 209 kJ energy, 3.1g protein, 1.7g fat, 4.6g carbohydrates, 3mg sodium, 200mg calcium, 7.5mg iron, 3mg zinc, 250μg RE vitamin A, 5μg vitamin D, 0.5mg vitamin B1, 0.5mg vitamin B2, 0.5μg vitamin B12, and 75μg folate. Intervention duration: 6 months, with 2 sachets per day. Produced by Tiantianai (Jiangsu) Biotechnology Co., Ltd., a certified supplier for maternal and child nutrition projects in China.The company has a Class D production workshop that meets the latest GMP standards for pharmaceuticals. The product has passed certifications for Food Safety Management System (ISO 22000) and Quality Management System (ISO 9001).
  Other Names: Yingyangbao
  Arms: Group 1; Group 2
Dietary Supplement: Probiotics — Dry, vacuum-sealed sachets containing white powder, odorless. Each 2g sachet contains 500*10^9 CFU of Lactobacillus plantarum LLY-606 and Pediococcus pentosaceus JQI-7. Intervention duration: 6 months, with 1 sachet per day. Produced by Jiangsu Wecare Biotechnology Co., Ltd., compliant with international standards (cGMP, FSSC 22000, HACCP, ISO 22000, ISO 9001).
  Arms: Group 1

SUMMARY:
The goal of this cluster randomized controlled trial is to study the effectiveness of the Nutrition Package (Yingyangbao) on improving malnutrition in children and adolescents aged 7-15 in Myanmar. The main questions it aims to answer are:

* What is the effectiveness of Nutrition Package intervention on the growth, development, and nutritional health of children and adolescents aged 7-15 in Myanmar?
* How safe and feasible is the Nutrition package? Researchers will compare the Nutrition Package plus probiotics, the Nutrition Package alone, and no intervention to see if the Nutrition Package improves malnutrition and other health outcomes of children and adolescents aged 7-15 in Myanmar.

Participants will receive Nutrition Package products for six months and have their height, weight, mid-upper arm circumference, and hemoglobin levels measured and compared at baseline and end.

DETAILED DESCRIPTION:
Study background:

Malnutrition among children and adolescents is a significant public health issue in developing countries, including Myanmar, severely affecting children and adolescents' growth, development, and overall health, and potentially leading to long-term adverse health outcomes or even death. Influenced by factors such as armed conflicts, the COVID-19 pandemic, and natural disasters, malnutrition in Myanmar has become even more pronounced.

Preliminary cross-sectional survey results indicate that the malnutrition rate among children and adolescents aged 7-15 in Special Region 4 of Myanmar is as high as 56.2%, with stunting, wasting (in children under 10), and underweight rates at 53.2%, 38.5%, and 5.0%, respectively. Additionally, health issues such as diarrhea, fever, skin and hair problems, and functional impairments are prevalent, with detection rates exceeding 40%. Analysis of influencing factors reveals that diet is a critical determinant of growth and development in this population. Nutrient assessments show insufficient daily intake of essential nutrients, including vitamin A, vitamin B1, vitamin B2, calcium, iron, and zinc. Children and adolescents aged 7-15 are in a critical period of growth and development, and nutrient deficiencies can lead to severe adverse health effects. Moreover, the prevalence of diseases such as diarrhea and fever may further impair nutrient absorption, creating a vicious cycle of malnutrition. Malnutrition among children and adolescents has become an urgent public health issue in Myanmar, necessitating interventions to improve these people's nutritional health.

Nutrition package, recommended by the WHO, has been proven effective in reducing the risks of anemia, stunting, underweight, and wasting in children under 5 in China. However, there is limited evidence on its effectiveness for older children and adolescents. Expert discussions have concluded that the current nutrition package formula, administered at a dose of two sachets per day, can meet the average nutrient requirements for different genders and age groups without exceeding the tolerable upper intake levels. The addition of probiotics to the nutrition packages may further enhance nutrient absorption, boost immune function, and reduce gastrointestinal diseases. The prior survey results indicate that children and adolescents in Special Region 4 of Myanmar currently do not have access to nutritional supplements, yet 98% of participants reported acceptance after using the nutrition package products. Therefore, implementing these nutritional interventions in this region might be safe, cost-effective, and feasible.

Based on the above facts, this study aims to conduct a pilot intervention using nutrition package among children and adolescents aged 7-15 in Special Region 4 of Myanmar. The goal is to evaluate the effectiveness and safety of these packages in improving the nutritional health of this population, providing essential scientific data to further enhance the growth, development, and nutritional health of children and adolescents in Myanmar.

Implementation Process:

Participants will be randomly assigned to two intervention groups or a control group. After the study, the control group will receive the most effective intervention for 3 months.

Sample size:

The sample size was calculated using the following formula:

N=(Zα/2+Zβ)^2×[p1(1-p1)+p0(1-p0)]/(p1-p0)^2 Based on the preliminary cross-sectional survey data, the stunting rate among children aged 7-15 in Myanmar is p0=53.2%. Assuming a reduction to p1=31.9% (RR = 0.60) after intervention, with α=0.025 and 1-β=0.9, the required sample size per group is 127. This study plans to enroll 200 participants per group to ensure adequate power.

Recruitment Process:

Target population and site: The study will be conducted at a primary school, with informed consent obtained from participants and the guardians.

Training: Surveyors from Health Poverty Action (HPA) will receive rigorous training.

Screening and informed consent: Eligible participants will be screened, and detailed study information will be provided to ensure informed consent.

Ethical approval: The study has been approved by the ethics committee of Tsinghua University and agreed by the Health Bureau of the Special Region 4, Eastern Shan State of Myanmar.

Data collection:

This cluster randomized controlled trial will collect baseline data through a structural questionnaire. Physical examinations will be taken at baseline and end. Collection of fecal samples will be taken at the ending of intervention. Adherence to the intervention and adverse events will be recorded to evaluate the effectiveness and safety of interventions.

Measurement:

1. Baseline characteristics: Demographics, medical history, lifestyle habits, and dietary intake.
2. Adherence: Distribution and adherence rates, recorded through returned packaging and usage logs.
3. Effectiveness:

   3.1. Anthropometric measurements: height, weight, mid-upper arm circumference. 3.2. Hemoglobin levels: measured using a HemoCue hemoglobin analyzer. 3.3. Fecal microbiota and parasites: analyzed from stool samples.
4. Safety: Adverse events will be recorded and monitored.

Potential Adverse Reactions:

Previous clinical applications have shown that nutrition packages and probiotics may cause adverse reactions, including systemic infections, harmful metabolic activities, excessive immune stimulation, gene transfer, and gastrointestinal discomfort. Individuals with severe gut microbiota imbalances may experience short-term abdominal pain or diarrhea after consumption.

Mitigation Measures:

A 7-day trial intervention will be conducted before the formal study begins. If a participant exhibits allergic reactions, gastrointestinal discomfort, or other symptoms deemed by a physician to be related to the nutrition package or probiotics, this participant will be excluded from the study. If a participant experiences adverse reactions during the formal intervention period, as determined by a physician, the participation in the study will be immediately terminated. In rare cases where symptoms persist after discontinuation, the research team, HPA, and the collaborating school will jointly provide follow-up treatment. The costs of such treatment will be covered by the research project.

Adverse Events and Special Protections:

Adverse events, including gastrointestinal discomfort, will be monitored and managed.

Special protections for children and adolescents include informed consent, free medical care for study-related injuries, and compensation if applicable.

This study aims to provide evidence on the effectiveness and safety of nutrition packages in improving the nutritional health of children and adolescents in Myanmar, contributing to public health interventions in the region.

Statistical Analysis:

Data will be analyzed using R software. Descriptive statistics, hypothesis testing, and regression analysis will be performed.

Quality Control:

Regular monitoring and follow-up will ensure data accuracy and participant safety. Biological samples will be anonymized and securely stored, with destruction after one year.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged 7-15 years.
2. Residing in the local area for more than 1 year.

Exclusion Criteria:

1. Individuals with severe metabolic diseases.
2. Diagnosed with HIV/AIDS.
3. Individuals with physical disabilities.
4. Individuals with severe mental conditions that may hinder their ability to cooperate with the study.
5. Those who have received other nutritional supplementation packages or fortified foods in the past 6 months.
6. Individuals with a history of intestinal diseases, other severe digestive system disorders, or metabolic disorders.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Physical examination | At the enrollment, later 3 month and later 6 month.
  Height and weight are measured using a height and weight meter, and mid-upper arm circumference is measured using an arm circumference ruler.

SECONDARY OUTCOMES:
Hemoglobin determination | At the enrollment, later 3 month and later 6 month.
  Hemoglobin of finger-tip blood is measured using a HemoCue hemoglobin analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Zhao, Principal Investigator — Vanke School of Public Health, Tsinghua University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Z, Li X, Sudfeld CR, Liu Y, Tang K, Huang Y, Fawzi W. The Effect of the Yingyangbao Complementary Food Supplement on the Nutritional Status of Infants and Children: A Systematic Review and Meta-Analysis. Nutrients. 2019 Oct 8;11(10):2404. doi: 10.3390/nu11102404. PMID 31597360